CLINICAL TRIAL: NCT02510612
Title: Perioperative Dexmedetomidine Affect Diabetic Patient's Glucose Metabolism
Brief Title: Dexmedetomidine Affect Diabetic Patient's Glucose Metabolism
Acronym: dadpgm
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaanxi Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Song yulong, Anesthetist, Shaanxi Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20150618
Record Dates: First submitted 2015-07-23; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes
Keywords: Dexmedetomidine; Diabetic; glycometabolism; sedation
MeSH Terms: conditions — Diabetes Mellitus | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Patients in group D will be given dexmedetomidine during anesthesia induction and maintenance phase respectively.In induction phase infuse 1μg/Kg of dexmedetomidine in 10 minutes， the speed in maintenance phase is 0.4μg/Kg.h
  Interventions: Drug: Dexmedetomidine
- placebo (Placebo Comparator): Patients in group P will be given normal saline during anesthesia induction and maintenance phase
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dexmedetomidine — During anesthesia induction, all patients will be given propofol,fentanyl,vecuronium bromide.But before induction start in Dexmedetomidine(D) group, patient will be given dexmedetomidine 1μg/Kg for 10 minutes In anesthesia maintenance, D group will be given dexmedetomidine 0.4μg/Kg.h until 40 minutes before the end of surgery
  Other Names: Yi Si
  Arms: Dexmedetomidine
Drug: placebo — During anesthesia induction, all patients will be given propofol,fentanyl,vecuronium bromide.But before induction start in Placebo(P) group, patient will be given placebo for 10 minutes In anesthesia maintenance, D group will be given placebo until 40 minutes before the end of surgery
  Other Names: normal saline
  Arms: placebo

SUMMARY:
Dexmedetomidine's Sedative Effect on Diabetic Patient

DETAILED DESCRIPTION:
Dexmedetomidine is a high selective α2 agonist,its sedative and analgesia feature is acclaimed. The pathogenesis of type 2 diabetes mellitus is associated with α2 excessive adrenaline receptors expression. This study is to evaluate whether the use of dexmedetomidine is helpful to Diabetic Patient through its antisympathetic effect

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 60
* Selective epigastrium surgery
* In

Exclusion Criteria:

* American Society of Anesthesiology (ASA) Physical Status>3
* Duration of operation >3 hours
* Hypovolemia,sinus bradycardia,atrioventricular block,severe hepatic and renal dysfunction,severe cardiac insufficiency

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
sedation level | from 5 minutes before medication to 10 minutes after Dexmedetomidine discontinuance，length of time frame is about 2 hours
  Ramsay score and BIS will be recorded before medication,5 min after medication, medication ending, 5 and 10 min after medication

SECONDARY OUTCOMES:
Heart rate | participants will be followed from operation day to first postoperative day，an expected average of 2 days
  recorded at before medication,5 min after medication, medication ending, 5 and 10 min after medication, before intubation, after intubation, after skin incision,60 minutes after skin incision, after extubation,first day after operation
Mean arterial pressure | participants will be followed from operation day to first postoperative day，an expected average of 2 days
  10 min after medication, before intubation, after intubation, after skin incision,60 minutes after skin incision, after extubation,first day after operation
blood glucose measured by Biochemical test | participants will be followed from operation day to first postoperative day，an expected average of 2 days
  it will be recorded immediately after the entrance to the operating room, before operation, 60 minutes after incision, after extubation, first day after operation
cortisol measured by Biochemical test | participants will be followed from operation day to first postoperative day，an expected average of 2 days
  it will be recorded immediately after the entrance to the operating room, before operation, 60 minutes after incision, after extubation, first day after operation
insulin measured by Biochemical test | participants will be followed from operation day to first postoperative day，an expected average of 2 days
  it will be recorded immediately after the entrance to the operating room, before operation, 60 minutes after incision, after extubation, first day after operation
adrenaline measured by Biochemical test | participants will be followed from operation day to first postoperative day，an expected average of 2 days
  it will be recorded immediately after the entrance to the operating room, before operation, 60 minutes after incision, after extubation, first day after operation
noradrenaline measured by Biochemical test | participants will be followed from operation day to first postoperative day，an expected average of 2 days
  it will be recorded immediately after the entrance to the operating room, before operation, 60 minutes after incision, after extubation, first day after operation